CLINICAL TRIAL: NCT03186586
Title: Ulipristal Versus Placebo for Women With Bleeding Induced by Mirena, a Randomized Clinical Trial
Brief Title: Ulipristal Versus Placebo for Women With Bleeding Induced by Mirena
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Luis Bahamondes, Professor of Gynecology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEMICAMP
Record Dates: First submitted 2016-12-12; First posted 2017-06-14 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Heavy Menstrual Bleeding; Abnormal Bleeding
Keywords: Heavy Menstrual Bleeding; Levonorgestrel relesing intrauterine system
MeSH Terms: conditions — Menorrhagia; Hemostatic Disorders | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulipristal acetate 5mg/day/five days (Experimental): Women with abnormal bleeding during use of Mirena will allocate to UPA or placebo Ulipristal acetate at 5mg/day/five days Ulipristal 5mg daily for 5 days at the bleeding episode
  Interventions: Drug: Ulipristal acetate
- Placebo 1 pill/day/five days (Placebo Comparator): Women with abnormal bleeding during use of Mirena will allocate to UPA or placebo Placebo at 1pill/day/five days Placebo one pill a day for 5 days at the bleeding episode
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulipristal acetate — 5mg/day/five days
  Arms: Ulipristal acetate 5mg/day/five days
Drug: Placebo — Placebo one pill a day for 5 days at the bleeding episode
  Arms: Placebo 1 pill/day/five days

SUMMARY:
Objectives: To assess if the administration of ulipristal acetate (UPA) in users of the levonorgestrel-releasing intrauterine system (LNG-IUS) with breakdown bleeding or abnormal bleeding, could be able to inhibit the bleeding and if this effect will be sustainable up to three months after treatment.

Material and methods: A total of 32 women aged between 18-45 years, users of the LNG-IUS with breakdown bleeding, abnormal bleeding or prolonged bleeding (bleeding more than 14 days) or episodes of bleeding with intervals less than 24 days). The study is an experimental, double blind randomized (16 women will receive UPA 5 mg/day/5 days; 16 women will receive placebo/1 time/day/5 day). The women will invited to participated at the Family Planning clinic at the day they consulted with the complaint of bleeding. That day they will allocated at random to UPA or placebo group. They will oriented to fill out a bleeding calendar through 90 days after the pill intake. In addition a ultrasonography scan will be perform before the first day of pill intake and at 90 days after.

Statistical analysis: A a pilot study the sample was estimated in 26 women (13 at each group) based at the estimative of success of 0.95 with UPA and 0.35 with placebo with significance of 0.05 and power of 80%. The sociodemographic characteristics will be analyzed as mean and SD and will compared through Mann-Whitney, Yates χ2 and Fisher exact tests as apropriate. Also, a regression analysis (Poisson analysis) with the dependent significant variables. The established level of significance will be p < 0.05.

DETAILED DESCRIPTION:
The LNG-IUS is a contraceptive method with high efficacy, long acting, reversible with contraceptive failure between 0.1 and 0.5/100 women/year. It released 20 mcg/day of LNG with a life span duration of 5 years. LNG is a synthetic progestin, 19-northestosterone, six times more potent than progesterone, with androgenic properties and with binding with sexual hormones, receptors of human steroids, including receptors of glucocorticoids and mineralocorticoids, with minimal capacity of binding with estrogen receptors. At endometrium level it induce antiproliferative effect and strong expression of local markers and endometrial decidualization, including the prolactin receptor and insulin-like growth factor. The mechanism of action includes effect upon cervical mucus which affects the sperm movements through the reproductive tract which affects fertilization. In some women could be ovulation inhibition. One of the main reason for discontinuation is breakdown bleeding, increase bleeding or abnormal bleeding including heavy menstrual bleeding (HMB) and spotting which is common at the first six month of use. Despite the fact that it is the main cause of discontinuation, there is no effective treatment for these cases. An effective treatment could help in the reduction of reduce the rates of discontinuation, improved the cost-effectiveness and quality of life of users.

A selective progesterone receptor modulator (SPRM) is Ulipristal Acetate (UPA) is approved in the European Union as Esmya® as a tretament to reduce the ueterine leiomyomas at te dose of 5 mg/day and it under evaluation at the dose of 5-10 mg as oral contraceptive.

This could be an option of treatment for HMB or abnormal bleeding induced by the LNG-IUS. UPA is agonist/antagonist and binding with progesterone to the receptor level. It has ovarian and endometrial activity, with dose-dependent effect in inhibition of ovulation and maturation of the endometrium. There are restricted evidences, that the administration of UPA induce a quick endometrial atrophy and stop the abnormal bleeding.

ELIGIBILITY:
Inclusion Criteria:

Women with complaints of abnormal bleeding during use of Mirena independently of the length of use

Exclusion Criteria:

Delivery in the last six months Breastfeeding Hematological disorder Use of anticoagulants Uterine leiomioma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Uterine bleeding control (stop bleeding) | Three months
  Uterine bleeding control (stop bleeding) among users of Mirena after use of UPA or placebo

SECONDARY OUTCOMES:
Endometrial control | Three months
  Endometrial thickness

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fava M, Peloggia A, Baccaro LF, Castro S, Carvalho N, Bahamondes L. A randomized controlled pilot study of ulipristal acetate for abnormal bleeding among women using the 52-mg levonorgestrel intrauterine system. Int J Gynaecol Obstet. 2020 Apr;149(1):10-15. doi: 10.1002/ijgo.13068. Epub 2019 Dec 11. PMID 31777949